CLINICAL TRIAL: NCT01774097
Title: Clinical and MR Imaging Assessments in Patients With Intermittent Claudication Following Injection of Bone Marrow Derived ALDH Bright Cells
Brief Title: Patients With Intermittent Claudication Injected With ALDH Bright Cells
Acronym: PACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Aldagen (Industry); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Dr Lemuel A Moye III, Professor - School of Public Health, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-SPH-12-0785; UM1HL087318-06 (NIH)
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
Keywords: Peripheral Artery Disease; Intermittent Claudication; Autologous Stem Cells; ALDH cells; Claudicants; PAD; Peak Walking Time; MRI; Vascular Flow; Anatomy; Perfusion
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALD-301 (Experimental): Participants will receive ALD-301 via intramuscular injection
  Interventions: Biological: ALD-301
- Placebo (vehicle) (Placebo Comparator): Participants will receive placebo (vehicle)via intramuscular injection
  Interventions: Biological: Placebo (vehicle)

INTERVENTIONS:
Biological: ALD-301 — Ten 1ml injections of ALD-301 in the index calf and posterior, lower thigh
  Other Names: ALDH Bright Cells; ALDHbr; Aldehyde dehydrogenase-bright cells
  Arms: ALD-301
Biological: Placebo (vehicle) — Ten 1ml injections of placebo in the index calf and posterior, lower thigh
  Other Names: Placebo; Vehicle; HSA; Human Serum Albumin
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to find out if aldehyde dehydrogenase bright (ALDHbr) cells taken from a patient's bone marrow can be placed safely, via intramuscular injections, into their affected calf and lower thigh muscles and improve blood flow and/or peak walking time in patients experiencing pain associated with blocked blood vessels in the leg.

DETAILED DESCRIPTION:
Peripheral Artery Disease (PAD) occurs when arteries in the arms and legs (most often the legs) become narrowed by plaque. Because of this plaque, patients with PAD are also at increased risk for heart attacks and strokes. Those with PAD often have intermittent claudication (blockage of blood vessels in the leg). This blockage decreases blood flow to the leg muscles, which can cause pain in one or both legs during exercise (such as during walking). Intermittent means the pain comes and goes. Because PAD interferes with circulation, worsening of this condition can increase pain in the leg; sometimes even during periods of rest.

Bone marrow contains special stem cells that may promote blood vessel growth, prevent cell death, and transform themselves into a number of tissues including new muscle. There is a small subpopulation of bone marrow mononuclear cells, called aldehyde dehydrogenase-bright (ALDHbr) cells, that is highly enriched in these types of stem cells. The enzyme in ALDHbr cells responds to damage signals and may play an important role in tissue repair.

In this study we investigate the safety and efficacy of bone marrow derived stem cells with particular characteristics in PAD patients with intermittent claudication and explore new end-points to evaluate therapeutic effects using novel MRI imaging modalities as well as traditional endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atherosclerotic peripheral artery disease with classic claudication (exercise-induced pain, cramps, fatigue, or other equivalent discomfort involving large muscle groups of the leg(s) that is consistently relieved by rest) or atypical leg pain (exertional leg pain that does not begin at rest or does not resolve consistently with rest) as defined by the San Diego Claudication Questionnaire.
2. Age ≥40 years
3. Resting ankle-brachial index <0.90 or a resting toe-brachial index of <0.70 at baseline testing
4. Presence of significant stenosis or occlusion of infrainguinal arteries including the superficial femoral artery, popliteal artery and/or infrapopliteal arteries as determined by: Duplex ultrasound imaging (occlusion or focal doubling of peak systolic velocity of one or more affected segments) OR lower extremity computed Tomography Angiography (CTA) OR lower extremity magnetic resonance angiography (MRA) OR lower extremity catheter-based contrast arteriography. Each of these noninvasive and invasive anatomic assessments will identify patients with at least a 50% stenosis in the affected segment.

Exclusion Criteria:

1. Presence of any musculoskeletal disease, cardiac or pulmonary disease, or neurological disease that limits the patient's ability to walk to fulfill protocol requirements (claudication must be the consistent primary exercise limitation)
2. Inability to complete treadmill testing per protocol requirements.
3. Ability to walk for more than 12 minutes on the treadmill during treadmill testing.
4. Patients who identify both legs as equivocally symptomatic or alternate between symptomatic legs on the baseline treadmill tests.
5. Patients with critical limb ischemia (ischemic rest pain or ischemia-related non healing wounds or tissue loss (Rutherford categories 4-6).
6. Recent (<3 months) infrainguinal revascularization (surgery or endovascular revascularization) or revascularization planned during study period
7. Patients with a patent infrainguinal bypass graft in the index limb, with or without evidence of a hemodynamically significant stenosis or other defect (kinking, pseudoaneurysm, or fistula). Patients with an occluded infrainguinal bypass graft or a patent aortobifemoral or femoral-femoral bypass graft are NOT excluded.
8. Patients with >2+ lower extremity pitting edema
9. Patients with myelodysplastic syndrome (MDS)
10. Patients who are pregnant or lactating, planning to become pregnant in the next 12 months, or are unwilling to use acceptable forms of birth control during study participation.
11. Congestive Heart Failure hospitalization within the last 1 month prior to enrollment
12. Acute coronary syndrome in the last 1 month prior to enrollment
13. Human Immunodeficiency Virus positive, active Hepatitis B Virus or Hepatitis C Virus Disease
14. History of cancer within the last 5 years, except basal cell skin carcinoma
15. Any bleeding diathesis defined as an International Normalized Ratio ≥ 2.0 (off anticoagulation therapy) or history of platelet count less than 100,000 or hemophilia
16. Contraindication to magnetic resonance imaging (MRI) (including knee/tibial/fibular replacement hardware in the index leg) or known allergy to MRI contrast media
17. Chronic kidney disease [effective Glomerular Filtration Rate <30 by modification of diet in renal disease (MDRD) or Mayo or Cockcroft-Gault formula]
18. Uncontrolled diabetes [Hemoglobin A1C (HbA1C)>8.5]
19. Planned change to (initiate or terminate) active involvement in a supervised exercise program (e.g., with a trainer, exercise protocol, and goals, such as in a peripheral arterial disease, cardiac or pulmonary rehabilitation program) during study participation
20. Plans to change medical therapy during the duration of the study, (i.e. patients who use cilostazol should remain on a stable dose for four weeks prior to enrollment and should not change doses for the 6 months of the study duration.) As always, cilostazol can be discontinued if new heart failure or intolerance occurs during study participation.
21. Any condition requiring immunosuppressant medications (e.g., for treatment of organ transplants, psoriasis, Crohn's disease, alopecia areata).
22. History of inflammatory or progressively fibrotic conditions (e.g. rheumatoid arthritis, systemic lupus erythematosis, vasculitic disorders, idiopathic pulmonary fibrosis, retroperitoneal fibrosis).
23. Patients with any untreated stenosis > 70% of the distal aorta, common iliac, or external iliac arteries by CT, Angiography or MRI imaging will be excluded from enrollment (patients with previously successfully revascularized inflow stenoses may enroll in PACE). Subjects who were screen failures for a flow-limiting proximal lesion may be rescreened 3 months after successful angioplasty/stenting.
24. Inability to provide written informed consent due to cognitive or language barriers (interpreter permitted)
25. Concurrent enrollment in another clinical interventional investigative trial.
26. Presence of any clinical condition that in the opinion of the principal Investigator or the sponsor makes the patient not suitable to participate in the trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simari, MD, Study Chair — Cardiovascular Cell Therapy Research Network
Locations (9):
- United States (9):
  - Stanford University School of Medicine (Falk Cardiovascular Research Center), Stanford, California
  - University of Florida-Department of Medicine, Gainesville, Florida
  - University of Miami-Interdisciplinary Stem Cell Institute, Miami, Florida
  - Orlando Health Inc., Orlando, Florida
  - Indiana Center for Vascular Biology and Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Clinical and Translational Science Institute at University of Minnesota, Minneapolis, Minnesota
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Perin EC, Silva G, Gahremanpour A, Canales J, Zheng Y, Cabreira-Hansen MG, Mendelsohn F, Chronos N, Haley R, Willerson JT, Annex BH. A randomized, controlled study of autologous therapy with bone marrow-derived aldehyde dehydrogenase bright cells in patients with critical limb ischemia. Catheter Cardiovasc Interv. 2011 Dec 1;78(7):1060-7. doi: 10.1002/ccd.23066. Epub 2011 May 18. PMID 21594960
- [Background] Perin EC, Murphy M, Cooke JP, Moye L, Henry TD, Bettencourt J, Gahremanpour A, Leeper N, Anderson RD, Hiatt WR, Lima JA, Venkatesh B, Sayre SL, Vojvodic RW, Taylor DA, Ebert RF, Hirsch AT; Cardiovascular Cell Therapy Research Network. Rationale and design for PACE: patients with intermittent claudication injected with ALDH bright cells. Am Heart J. 2014 Nov;168(5):667-73. doi: 10.1016/j.ahj.2014.07.021. Epub 2014 Jul 30. PMID 25440794
- [Derived] Perin EC, Murphy MP, March KL, Bolli R, Loughran J, Yang PC, Leeper NJ, Dalman RL, Alexander J, Henry TD, Traverse JH, Pepine CJ, Anderson RD, Berceli S, Willerson JT, Muthupillai R, Gahremanpour A, Raveendran G, Velasquez O, Hare JM, Hernandez Schulman I, Kasi VS, Hiatt WR, Ambale-Venkatesh B, Lima JA, Taylor DA, Resende M, Gee AP, Durett AG, Bloom J, Richman S, G'Sell P, Williams S, Khan F, Gyang Ross E, Santoso MR, Goldman J, Leach D, Handberg E, Cheong B, Piece N, DiFede D, Bruhn-Ding B, Caldwell E, Bettencourt J, Lai D, Piller L, Simpson L, Cohen M, Sayre SL, Vojvodic RW, Moye L, Ebert RF, Simari RD, Hirsch AT; Cardiovascular Cell Therapy Research Network (CCTRN). Evaluation of Cell Therapy on Exercise Performance and Limb Perfusion in Peripheral Artery Disease: The CCTRN PACE Trial (Patients With Intermittent Claudication Injected With ALDH Bright Cells). Circulation. 2017 Apr 11;135(15):1417-1428. doi: 10.1161/CIRCULATIONAHA.116.025707. Epub 2017 Feb 16. PMID 28209728
- See also: Cardiovascular Cell Therapy Research Network — http://www.cctrn.org
- See also: National Heart, Lung, and Blood Institute — http://www.nhlbi.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at seven Network centers and their associated satellite facilities between 6/13/2013 and 12/8/2015. The main centers are located in Texas, Florida (2 locations), Minnesota, Kentucky, Indiana, and California. Study brochures, patient informational DVDs, and clinicaltrials.gov were among the tools used for recruitment.
Groups:
- ALDHbr: Participants will receive ALDHbr via intramuscular injection
  ALDHbr: Ten 1ml injections of ALDHbr in the index calf and posterior, lower thigh
- Placebo (Vehicle): Participants will receive placebo (vehicle) via intramuscular injection
  Placebo (vehicle): Ten 1ml injections of placebo in the index calf and posterior, lower thigh
Period: Overall Study
Arm/Group | ALDHbr | Placebo (Vehicle)
Started | 40 | 42
Completed | 38 | 40
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Information for 4 participants is not available due to patient withdrawal from the study.
Groups:
- ALDHbr: Participants will receive ALDHbr cells via intramuscular injection
  ALDHbr: Ten 1ml injections of ALDHbr cells in the index calf and posterior, lower thigh
- Total: Total of all reporting groups
Arm/Group | ALDHbr | Placebo (Vehicle) | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (8.6) | 66.2 (8.7) | 66.2 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 26 | 31 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Peak Walking Time (PWT)
Description: The placebo adjusted average change over time in the maximum time (in minutes) walked by a patient on a treadmill under standardized conditions. The patient continues the test until walking can no longer be tolerated because of claudication symptoms.
Time Frame: Assessed at baseline and 6 months
Population: Participants who had available analyzable baseline and 6 month treadmill test results.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 37 | 39
minutes | 2.2 (3.9) | 1.2 (2.7)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.238, t-test, 2 sided — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.6 to 2.5], Standard Error of Mean 0.8

2. Primary Outcome: Leg Collateral Count (Via Contrast Enhanced-MR)
Description: The placebo adjusted average change in the number of collateral vessels over time.
Time Frame: Assessed at baseline and 6 months
Population: Participants who had available analyzable baseline and 6 month MRI imaging
Measure: Mean (Standard Deviation); unit: vessel count
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 37 | 38
vessel count | 1.5 (2.7) | 0.6 (2.2)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.116, t-test, 2 sided — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.2 to 2.1], Standard Error of Mean 0.6

3. Primary Outcome: Peak Hyperemic Popliteal Flow (Phase Contrast MRA)
Description: The placebo adjusted average change in peak hyperemic popliteal flow (mL/s) over time.
Time Frame: Assessed at baseline and 6 months
Population: Participants who had available analyzable baseline and 6 month MRI imaging
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 35 | 36
ml/sec | 0.2 (1.5) | 0.2 (1.9)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.978, t-test, 2 sided — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.4

4. Primary Outcome: Capillary Perfusion
Description: The placebo adjusted average change in capillary perfusion over time.
Time Frame: Assessed at baseline and 6 months
Population: Participants with available analyzable MRI imaging at baseline and 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 38 | 38
percent | -0.42 (2.40) | -0.25 (2.36)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.752, t-test, 2 sided — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = -0.17, 95% CI 2-sided [-1.26 to 0.91], Standard Error of Mean 0.55

5. Secondary Outcome: Pre-exercise Ankle-Brachial Index (ABI)
Description: ABI is the ratio of the blood pressure at the ankle to the blood pressure of the upper arm. Pre-exercise ABI is collected routinely with the patient supine immediately prior to a treadmill test. This measure represents the placebo adjusted average change over time in arm and pedal (ankle) blood pressure. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 3mos, and 6 mos)
Population: Participants with available analyzable ABI data at baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 36 | 39
ratio | 0.61 (0.17) | 0.64 (0.14)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.871, Regression, Linear — Threshold 0.05; no adjustment for multiple comparisons per protocol; interaction term = 0.00, 95% CI 2-sided [-0.02 to 0.03], Standard Error of Mean 0.01

6. Secondary Outcome: Post-exercise Ankle-Brachial Index (ABI)
Description: ABI is the ratio of the blood pressure at the ankle to the blood pressure of the upper arm. Post-exercise ABI is collected routinely with the patient supine immediately following a treadmill test. This measure represents the placebo adjusted average change over time in arm and pedal (ankle) blood pressure. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 3mos, and 6 mos)
Population: Participants with available analyzable ABI at baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 36 | 39
ratio | 0.30 (0.15) | 0.34 (0.19)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.256, Regression, Linear — Threshold 0.05; no adjustment for multiple comparisons per protocol; interaction term = -0.02, 95% CI 2-sided [-0.06 to 0.02], Standard Error of Mean 0.02

7. Secondary Outcome: Claudication Onset Time (COT)
Description: Claudication Onset Time (COT) is the walking time at which patients first experience leg pain during a treadmill test. The measure represents placebo adjusted average change over time (in minutes) in the time walked by a patient on a treadmill under standardized conditions before the onset of claudication symptoms, regardless of whether this is manifested or characterized as muscle pain, ache, cramp, numbness or fatigue. This does not include joint pain or other pain not associated with claudication. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 3mos, and 6 mos)
Population: Participants who had available analyzable baseline, 3 month, and 6 month treadmill test results.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 34 | 35
minutes | 2.8 (1.9) | 2.5 (1.7)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.241, Regression, Linear; interaction term = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.2

8. Secondary Outcome: Peak Walking Time (PWT)
Description: The average change in maximum time (in minutes) walked by a patient on a treadmill under standardized conditions. The patient continues the test until walking can no longer be tolerated because of claudication symptoms.
Time Frame: Assessed at baseline and 3 months
Population: Participants who had available analyzable baseline, 3 month, and 6 month treadmill test results.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 36 | 38
minutes | 7.1 (4.4) | 6.0 (4.0)

9. Secondary Outcome: Peripheral Artery Questionnaire (PAQ)
Description: The Peripheral Artery Questionnaire (PAQ) assesses subjective physical limitations, leg symptoms, social function, treatment satisfaction, and quality of life. It is administered as a self report. Higher scores are indicative of better outcome. The summary scores is compiled by taking the mean of five subscales generated from the original questions. Range: Minimum score is 11.1, maximum 85. The measure represents placebo adjusted average change in Peripheral Artery Questionnaire (PAQ) summary score assessed over time. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 1mos, 3mos, and 6 mos)
Population: Participants who had available analyzable baseline, 1 month, 3 month, and 6 month PAQs.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 38 | 40
scores on a scale | 63.9 (21.5) | 55.2 (20.0)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.131, Regression, Linear — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = 2.1, 95% CI 2-sided [-0.6 to 4.8], Standard Error of Mean 1.4

10. Secondary Outcome: Walking Impairment Questionnaire (WIQ)-Walking Distance Score
Description: The Walking Impairment Questionnaire (WIQ) assesses the severity of the subjective walking impairment on distance, speed, and stair climbing scales. It is administered as a self report. Range: Minimum score is 0.2, maximum 100. The measure represents the placebo adjusted average change in WIQ walking distance score assessed over time. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 1mos, 3mos, and 6 mos)
Population: Participants who had available analyzable baseline, 1 month, 3 month, and 6 month WIQs.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 37 | 34
scores on a scale | 35.6 (30.1) | 23.0 (18.8)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.626, Regression, Linear — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = 0.9, 95% CI 2-sided [-2.6 to 4.2], Standard Error of Mean 1.7

11. Secondary Outcome: Walking Impairment Questionnaire (WIQ)- Walking Speed Score
Description: The Walking Impairment Questionnaire (WIQ) assesses the severity of the subjective walking impairment on distance, speed, and stair climbing scales. It is administered as a self report. Range: Minimum score is 0, maximum 87. The measure represents the placebo adjusted average change in WIQ walking speed score assessed over time. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 1mos, 3mos, and 6 mos)
Population: Participants who had available analyzable baseline, 1 month, 3 month, and 6 month WIQs
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 35 | 37
scores on a scale | 48.9 (20.7) | 41.8 (25.1)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.591, Regression, Linear — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = -0.9, 95% CI 2-sided [-4.1 to 2.3], Standard Error of Mean 1.6

12. Secondary Outcome: Walking Impairment Questionnaire (WIQ)-Ability to Climb Stairs Score
Description: The Walking Impairment Questionnaire (WIQ) assesses the severity of the subjective walking impairment on distance, speed, and stair climbing scales. It is administered as a self report. Range: Minimum score is 0, maximum 100. The measure represents the placebo adjusted average change in WIQ ability to climb stairs score assessed over time. The reported value is the estimate from regression analysis of the slope of the placebo adjusted measure over the time course of the trial adjusted for baseline weight.
Time Frame: Assessed as a trajectory (baseline, 1mos, 3mos, and 6 mos)
Population: Participants who had available analyzable baseline, 1 month, 3 month, and 6 month WIQs
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ALDHbr | Placebo (Vehicle)
Number analyzed (Participants) | 35 | 38
scores on a scale | 46.3 (29.9) | 43.8 (32.0)
Statistical Analysis 1: Comparison: ALDHbr vs Placebo (Vehicle); Test type: Superiority or Other; p = 0.722, Regression, Linear — Threshold 0.05; no adjustment for multiple comparisons per protocol; Mean Difference (Net) = 0.7, 95% CI 2-sided [-3.3 to 4.7], Standard Error of Mean 2.0

ADVERSE EVENTS:
Time Frame: Events reported are from randomization date to the 6 month endpoint data collection window (i.e 210 days post intervention)
Description: Events were assessed systematically at each study visit during the physical exam assessment. A standard workbook was used to collect event details. Sponsor safety team reviewed events and requested additional documentation as needed.
Arm/Group | ALDHbr | Placebo (Vehicle)
Serious Adverse Events (participants affected / at risk) | 4/40 | 8/42
Other Adverse Events (participants affected / at risk) | 1/40 | 6/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALDHbr (N=40) | Placebo (Vehicle) (N=42)
Acute Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Anginal discomfort (symptomatic) (Cardiac disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Compression of fractured vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hematoma (left popliteal) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CABG (Surgical and medical procedures) | 0 (0) | 1 (1)
Ischemic limb pain (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial disease (worsening) (Vascular disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALDHbr (N=40) | Placebo (Vehicle) (N=42)
Facial paralysis (Bell's palsy) (Nervous system disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 2 (2)
Post operative hip pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size. Only follow up to 6 months. Limitation in the cell dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes